CLINICAL TRIAL: NCT01724073
Title: Effect of the Regular Consumption of Leafy-vegetable Sauces, Rich in Iron, Zinc and Vitamin A, on Growth and Micro-nutrient Status of Young Children in Burkina Faso
Brief Title: Regular Consumption of Leafy Vegetable Sauces and Micro-nutrient Status of Young Children in Burkina Faso
Acronym: Instapa-WP4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Approval denied by national ethical committee of Burkina Faso
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: IRSAT DTA Burkina Faso (Unknown); Hopital Yalgado Ouedraogo Burkina Faso (Unknown)
Responsible Party: Principal Investigator, Claire Mouquet-Rivier, PhD, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRD-UMR204-NA1; IRSAT-DTA Burkina Faso (Other: research institute)
Record Dates: First submitted 2012-10-25; First posted 2012-11-09 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Anemia
Keywords: food to food fortification strategy; leafy vegetable; iron; zinc; vitamin A; growth
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Leafy vegetable-fish sauce (Experimental): one meal per day, 6 days a week, with leafy vegetable-fish sauce + tô, a local cereal-based paste
  Interventions: Dietary Supplement: Leafy vegetable-fish sauce
- Leafy vegetable-fish/liver sauce (Experimental): one meal per day, 6 days a week, 5 days with leafy vegetable-fish sauce + tô, 1 day with leafy vegetable-liver sauce + tô
  Interventions: Dietary Supplement: Leafy vegetable-fish/liver sauce
- Misola (Experimental): one meal per day, 6 days a week, with gruel prepared with the fortified Misola flour
  Interventions: Dietary Supplement: Misola
- no test food (No Intervention): control group receiving no test food

INTERVENTIONS:
Dietary Supplement: Leafy vegetable-fish sauce
  Arms: Leafy vegetable-fish sauce
Dietary Supplement: Leafy vegetable-fish/liver sauce
  Arms: Leafy vegetable-fish/liver sauce
Dietary Supplement: Misola
  Arms: Misola

SUMMARY:
A food-to-food fortification strategy has been designed based on traditional foods of Burkina Faso to fight against micronutrient deficiencies in young children. Leafy vegetable sauces were formulated to improve their micronutrient contents and bioavailability. This efficacy study was designed to assess the effects of the regular consumption (one meal per day, 6 days per week) of these leafy-vegetable sauces enriched or not with liver on iron, zinc and vitamin A status, growth and morbidity of young children from poor urban districts of Ouagadougou. The study is conducted by IRD and IRSAT-DTA and will last 6 months. 432 12-15 month-old children will be recruited and randomly assigned to one of the four following arms: three intervention groups, the two first receiving leafy vegetable sauce, the third one receiving one meal made of the fortified Misola gruel. In these three arms, blood samples will be collected at the beginning and at the end of the study. The fourth arm is an external control group and will not receive any food. In this fourth arm, blood samples will be collected only at the end of the study. Biochemical indicators of micronutrient status will be determined, and anthropometric data will be collected in all children. Morbidity will also be assessed in children of intervention groups.

DETAILED DESCRIPTION:
Micronutrient deficiencies and stunting are a major health concern in young children of many developing countries, including Burkina Faso. This poor nutritional status affects health, with a much higher risk for mortality, and delayed physical and cognitive development.

The INSTAPA project focuses on the improvement of millet-, sorghum-, maize-, and cassava-based foods for young children in sub-Saharan Africa to safely prevent deficiencies of iron, zinc, and vitamin A.

Food-to-food fortification strategy has rarely been tested in efficacy studies, despite its promising sustainability. The study will be conducted by IRD, IRSAT-DTA, with funding of the European Union.

Subjects of the study, 12-15 month old burkinabè children will be divided into 4 arms. 108 children per group (432, in all) will be recruited in order to have 90 children in each group after exclusion due severe anemia or hemoglobinopathy. Each enrolled child will be dewormed according to WHO recommendations, and receive a bed-net for malaria prevention.

Three of these four groups will receive one test meal per day, 6 days per week (except Sunday)in canteens located in study districts. Investigators will record every day the amount of food consumed and morbidity in each child.

* one intervention group receiving leafy vegetable-fish sauce + cereal-based paste called tô,
* one intervention group receiving leafy vegetable-fish sauce + cereal-based paste called tô 5 days/week and leafy vegetable-fish sauce + tô 1 day/week,
* one 'positive control' group receiving a fortified gruel prepared from Misola Flour In these three arms, blood samples will be collected at the beginning and at the end of the study.

The fourth arm is an external control group and will not receive any food. In this fourth arm, blood samples will be collected only at the end of the study.

Biochemical indicators of iron, zinc and vitamin A status will be determined, and anthropometric data will be collected in all children.

The study is submitted to the Ethical committee of the Ministry of Health of Burkina Faso and to the review board of the local drug administration (DGPML) for approval, as well as to the Ethical committee of IRD (France).

According to the results, recommendations on the young child diet will be formulated for the attention of the staff of health facilities and families.

ELIGIBILITY:
Inclusion Criteria:

* age between 12 and 15 months
* signed informed consent by parent or caregiver
* accept to eat every ingredient used for the preparation of the sauces

Exclusion Criteria:

* any chronic illness affecting growth or iron status (thalassemia or sickle-cell anemia) no informed consent
* severe acute malnutrition which will require direct treatment
* severe anemia which will require direct treatment

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Change in micronutrient status | six months
  iron, zinc and vitamin A status using plasma concentrations
Growth | 6 months
  Weight, length, mid-upper arm circumference

SECONDARY OUTCOMES:
food consumption | at t=around 1 month
  weighed record during one whole day
Intake of experimental food | up to 6 months
  the amount of experimental food eaten by each child will be weighed every day
Morbidity | up to 6 months
  daily record by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claire Mouquet-Rivier, PhD, Principal Investigator — Institut de Recherche pour le Developpement; Bréhima Diawara, PhD, Principal Investigator — Institut de Recherche en Sciences Aplliquées et Technologie - DTA
Locations (1):
- Institut de Recherche en Sciences Aplliquées et Technologie - DTA, Ouagadougou, Centre Region, Burkina Faso

REFERENCES:
- See also: The INSTAPA project receives funding from the European Union's Seventh Framework Programme [FP7/2007-2013] under grant agreement no 211484 — http://www.instapa.org/instapa